CLINICAL TRIAL: NCT07201922
Title: A Double Blind, Randomized, Placebo-controlled Exploratory Trial to Investigate the Efficacy and Safety of Nerandomilast Over 24 Months When Administered in Individuals With Interstitial Lung Abnormalities and a Family History of Pulmonary Fibrosis to Reduce the Risk of Worsening (DROP-FPF)
Brief Title: A Study to Test Whether Nerandomilast Can Help Slow Down Changes in the Lung in People With a Family History of Pulmonary Fibrosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1305-0069; 2025-522383-33 (Registry Identifier: CTIS); U1111-1322-6453 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-09-30; First posted 2025-10-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Familial Pulmonary Fibrosis; Interstitial Lung Abnormalities; Interstitial Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nerandomilast (Experimental)
  Interventions: Drug: Nerandomilast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nerandomilast — Nerandomilast
  Other Names: BI 1015550, JASCAYD®
  Arms: Nerandomilast
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to people aged 40 years or older who have at least 1 family member with pulmonary fibrosis. Pulmonary fibrosis is a condition where lung tissue becomes scarred, making it harder to breathe. People can join if a lung scan shows early changes in the lung, called interstitial lung abnormalities, which may lead to lung scarring. People with family members who have pulmonary fibrosis are more likely to develop it themselves. That is why it is important to check early for lung changes and find ways to prevent the condition from getting worse. The purpose of this study is to find out whether a medicine called nerandomilast can help slow down changes in the lung in people with a family history of pulmonary fibrosis.

Participants are put into one of 2 groups randomly, which means the group is chosen by chance. One group takes nerandomilast tablets, and the other group takes placebo tablets. Placebo tablets look like nerandomilast tablets but do not contain any medicine. Participants take a tablet twice a day for about 2 to 3 years. There is a 3 out of 5 chance that participants will receive nerandomilast instead of the placebo.

Participants are in the study for about 2 to 3 years. Participants visit the study site multiple times: more frequently during the first 2 years (about every 3 months), and then every 6 months thereafter. In the 3rd year, participants also have phone calls with the site staff every 3 months.

Doctors regularly test lung function and take chest scans to see if the treatment works. The results are compared between the 2 groups to see if nerandomilast helps. The doctors also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥40 years of age at the time of first signed informed consent at Visit 1a
* Participants must have at least 1 first-degree relative (biological parent, sibling, or child) with confirmed pulmonary fibrosis (idiopathic pulmonary fibrosis [IPF], idiopathic nonspecific interstitial pneumonia [NSIP], and/or pulmonary fibrosis due to known genetic cause [e.g. short telomere syndrome, mucin 5B (MUC5B) mutation, surfactant protein mutations])
* High resolution computed tomography (HRCT) scan with evidence of interstitial lung abnormalities involving at least 5% of a single lung zone or interstitial lung disease (ILD), based on central evaluation
* Forced vital capacity (FVC) ≥80% of predicted normal at Visit 1b
* Diffusing capacity of the lungs for carbon monoxide (DLCO) corrected for hemoglobin ≥70% of predicted normal at Visit 1b Further inclusion criteria apply.

Exclusion Criteria:

* Prior known pulmonary fibrosis that, in the opinion of the Investigator, requires treatment with approved therapies
* Prebronchodilator forced expiratory volume in 1 second (FEV1)/FVC <0.7 at Visit 1b
* HRCT findings consistent with probable or definite usual interstitial pneumonia (UIP) pattern
* Any medical condition that is known to predispose to the development of pulmonary fibrosis (e.g. known connective tissue disease)
* Prior or current use of nerandomilast, nintedanib, or pirfenidone Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-23 (Estimated)

PRIMARY OUTCOMES:
Time to physiologic or radiologic worsening of ILA/ILD over the whole trial | up to 164 weeks
  Defined as relative decline in forced vital capacity (FVC) % predicted of >10% from baseline; or absolute decline in diffusing capacity of the lungs for carbon monoxide (DLCO) % predicted >10% from baseline; or absolute increase in weighted reticulovascular score (wRVS) >2% and total disease extent (TDE) >2.5% on chest high resolution CT scan (HRCT), as measured by e-Lung Quantitative HRCT scoring, from baseline

SECONDARY OUTCOMES:
Absolute change from baseline in wRVS on e-Lung Quantitative HRCT scoring at weeks 26, 52, and 104 | at baseline, at weeks 26, 52 and 104
Absolute change from baseline in TDE on e-Lung Quantitative HRCT scoring at weeks 26, 52, and 104 | at baseline, at weeks 26, 52 and 104
Absolute change from baseline in FVC (% predicted) at weeks 26, 52, and 104 | at baseline, at weeks 26, 52 and 104
Absolute change from baseline in DLCO (% predicted) at weeks 26, 52, and 104 | at baseline, at weeks 26, 52 and 104
Time to relative decline from baseline in FVC (% predicted) of >10% over 52 weeks and over the whole trial | up to 164 weeks
Time to absolute decline from baseline in FVC (% predicted) of >5% over 52 weeks and over the whole trial | up to 164 weeks
Time to absolute decline from baseline in DLCO (% predicted) of >10% over 52 weeks and over the whole trial | up to 164 weeks
Time to absolute increase in wRVS >2% and TDE >2.5% on chest HRCT, as measured by e-lung quantitative HRCT scoring over 52 weeks and over the whole trial | up to 164 weeks
Time to physiologic or radiologic worsening of ILA/ILD over 52 weeks | up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (50):
- United States (12):
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Clinical Research Specialists LLC - Kissimmee, Kissimmee, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medicine-New York-60569, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (5):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - Hospital Italiano de Buenos Aires, CABA
  - Centro de Investigación Clinica Belgrano, CABA
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Consultorios Médicos del Buen Ayre, Capital Federal
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- France (5):
  - HOP Louis Pradel, Bron
  - INS Coeur Poumon, Lille
  - HOP Bichat, Paris
  - HOP Pontchaillou, Rennes
  - Hôpital Larrey - CHU de Toulouse, Toulouse
- Germany (4):
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Lungenfachklinik Immenhausen, Immenhausen
  - Krankenhaus Bethanien gGmbH, Solingen
- Italy (3):
  - IRCCS MultiMedica, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Japan (6):
  - Tosei General Hospital, Aichi, Seto
  - Tsuboi Hospital, Fukushima, Koriyama
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- South Korea (3):
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital de Galdakao, Galdakao
  - Hospital Universitari de Bellvitge, L'Hospitalet Del Llobregat
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Virgen del Rocío, Seville
- United Kingdom (2):
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency